CLINICAL TRIAL: NCT01216007
Title: A Pilot Study to Investigate Plasma Bupivacaine Concentrations in Children Receiving Total Intravenous Anaesthesia and Caudal Analgesia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Simon Whyte, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H10-01501
Record Dates: First submitted 2010-08-30; First posted 2010-10-07 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Anesthesia
Keywords: Plasma; bupivacaine; concentration; caudal; epidural; TIVA; Inhalational; anesthesia; Caudal epidural
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TIVA (Active Comparator): TIVA
  Interventions: Drug: propofol
- Inhalational (Active Comparator): Inhalational/volatile general anesthetic
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: propofol — In the TIVA group, IV access will be obtained as per BCCH routine, with caregiver present. 2% lidocaine 1 mg/kg will be administered via IV to prevent venous pain before induction of anaesthesia with propofol, as per BCCH standard. Induction of anaesthesia will be achieved with an IV bolus of propofol 5 mg/kg and remifentanil 2.5 mcg/kg. Anaesthesia will be maintained with an infusion of propofol 200-400 mcg/kg/min and remifentanil 0.1-0.2 mcg/kg/min. Once the subject is under general anaesthesia, the anaesthesiologist will place a second IV cannula, specifically for the collection of blood samples. This cannula will not be in the same limb as the propofol infusion.
  Arms: TIVA
Drug: sevoflurane — In the volatile anaesthesia group, induction of anaesthesia will be achieved with inhalation of sevoflurane (5-8% in O2/air). Maintenance of anaesthesia will continue with a volatile agent of the anaesthesiologist's choice.
  Arms: Inhalational

SUMMARY:
The objective of this pilot study is to compare plasma [bupivacaine] between two groups of paediatric patients under general anaesthesia who will all receive regional caudal anaesthesia with bupivacaine: group 1 will receive TIVA and group 2 will receive a volatile anaesthetic.

DETAILED DESCRIPTION:
Hypothesis:

The investigators hypothesize that there will be a detectable difference in free plasma [bupivacaine] between these two treatment groups, with lower free plasma [bupivacaine] in the TIVA group.

Background:

Local anesthetics (LA) are frequently administered intra-operatively, in combination with general anaesthesia, for pain management in children. Although highly effective in this regard, LAs possess a narrow margin of safety. High plasma levels can cause toxicity in both the central nervous system (CNS) and the cardiovascular system (CVS) and may result from either the correct placement of an excessive dose or an inadvertent intravenous (IV) injection of a correct dose.

Specific Objectives:

The objective of this pilot study is to compare plasma [bupivacaine] between two groups of paediatric patients under general anaesthesia who will all receive regional caudal anaesthesia with bupivacaine: group 1 will receive TIVA and group 2 will receive a volatile anaesthetic.

Methods:

Induction of anesthesia: The TIVA group will receive the BCCH standard regimen comprising induction with propofol 5 mg/kg and remifentanil 2.5 mcg/kg, followed by maintenance infusion of propofol 200-400 mcg/kg/min and remifentanil 0.1-0.2 mcg/kg/min. Total cumulative Intralipid® doses will be recorded at times of caudal injection and blood sampling. The volatile anesthesia group will undergo inhalational induction with sevoflurane in oxygen, followed by maintenance with a volatile agent of the anesthesiologist's choice. In both groups, airway management will be at the discretion of the anesthesiologist. Standard minimum monitoring will be applied. A caudal epidural will then be performed using a standard technique.

Administration of caudal analgesia and whole blood sampling: A caudal dose of 1 ml/kg of 0.25% bupivacaine (2.5 mg/kg) with 1 in 200 000 epinephrine will be administered at time zero (T0). Venous blood samples of 5 ml will be obtained from a second indwelling IV cannula 15 (T1) and 30 (T2) min after caudal injection. These will be collected into EDTA-containing tubes by the PART research assistant and transferred to the BCCH pharmacy research technician (blinded to anesthetic technique) for analysis. Blood samples will be immediately centrifuged. The extracted plasma will be frozen at -850C. Total and free bupivacaine plasma concentrations will be determined using high-pressure liquid chromatography (HPLC) and ultrafiltration.

Data Analysis:

This pilot study will have two primary outcome measures, total and free plasma bupivacaine concentrations. These data will be presented as mean (± SD) at T1 and T2. Normal distribution will be tested by histogram plot. Between-group (TIVA vs. volatile anaesthesia) comparisons of total and free plasma bupivacaine levels will be performed using appropriate analyses of variance. This analysis will determine if there is a detectable difference in plasma concentrations between the TIVA and volatile anaesthesia groups. These data will then be used in a power calculation to determine necessary group sizes for a future randomized controlled trial (RCT) study. Statistical analysis will be conducted using Analyse-It® (Analyse-It Software, Leeds, UK) in consultation with a statistician (Clinical Research Statistical Unit).

ELIGIBILITY:
Inclusion criteria:

* Age 6 months - 5 years
* ASA I-II
* Undergoing elective day surgery for which combined general and caudal epidural anaesthesia is indicated
* Written parental/guardian informed consent

Exclusion criteria:

* Weight and body mass index < 3rd or > 97th percentile for age
* Any contraindication to caudal injection
* Renal, hepatic, neuromuscular or cardiac disease
* Acute inflammatory process or infectious processes that provoke an acute phase response, ongoing or resolved less than 2 weeks prior to recruitment day (such as recent surgery, respiratory tract infection (including colds), urinary tract infection, infectious or inflammatory gastroenteritis, otitis media, skin or wound infection, cholecystitis, pancreatitis, hepatitis, meningitis) Chronic co-existing inflammatory diseases (eg, inflammatory bowel disease, juvenile arthritis, cystic fibrosis, autoimmune disease, connective tissue disease, chronic liver disease)

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Total and free plasma bupivacaine concentrations
  5 mL blood sample will be obtained at 15 and 30min. Total and free plasma bupivacaine concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Simon Whyte, Dr., Principal Investigator — The University of British Columbia
Locations (1):
- BC Children's Hospital, Department of Anesthesia, Vancouver, British Columbia, Canada